CLINICAL TRIAL: NCT03071705
Title: Effect of Metformin in Combination With Tyrosine Kinase Inhibitors (TKI) on Clinical, Biochemical and Nutritional in Patients With Non-Small Cell Lung Carcinoma (NSCLC): Randomized Clinical Trial
Brief Title: Metformin Plus TKI Use in Patients With Non-Small Cell Lung Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, Head Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 016/018/ICI; Ethics Committe (Other: CEI/1019/16)
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Adenocarcinoma; Tyrosine Kinase Mutation; EGFR Gene Mutation
Keywords: NSCLC; metformin; metformin plus TKI; EGFR positive status
MeSH Terms: interventions — Metformin; Erlotinib Hydrochloride; Afatinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): TKI plus Metformin
  Interventions: Drug: Metformin; Drug: TKI
- Control (Active Comparator): TKI
  Interventions: Drug: TKI

INTERVENTIONS:
Drug: Metformin — 500 mg PO BID
  Other Names: DABEXR
  Arms: Intervention
Drug: TKI — standard dose
  Other Names: erlotinib; afatinib; gefitinib

SUMMARY:
Treatment for patients with mutation in the epidermal growth factor receptor (EGFR) with specific domain tyrosine kinase inhibitors (TKIs) has given place to objective clinical response, increase in progression-free survival (PFS) compared to cytotoxic chemotherapy. However, despite clinical success with different TKIs, most patients eventually develop acquired resistance to these agents after an average period of time of 10 months.

Recently metformin, an oral hypoglycemic agent, has been associated with reduction in the global risk of incidence and mortality of different types of cancer, by exercising anti-tumor properties. Its role as a chemo-preventive and adjuvant drug in overcoming acquired resistance to chemotherapy, target therapy and immunotherapy in NSCLC is still under discussion.

However, preclinical data support the role as an adjuvant drug in the treatment of NSCLC in combination with chemotherapy or EGFR-TKIs. This evidence led to examine the effects of metformin in combination with EGFR-TKIs in a NSCLC cellular line panel, obtaining a different sensibility to the unique use with EGFR-TKIs. The combination of metformin and TKIs reduced the colony forming capacity and proliferation, and induced a huge pro-apoptotic effect in NSCLC cellular lines and resistance in EGFR-TKIs. This suggests that metformin may reduce the resistance to TKIs. A retrospective study in patients from our institution from 2008 to 2014, showed significant clinical benefit in patients who used metformin, improving the global survival. Based on these considerations, we propose a phase II randomized study to assess the effect and safety of metformin in combination with TKIs as second line therapy in patients with NSCLC in advanced stages with EGFR mutation.

The main objective of this study is to assess the progression-free survival period in patients with advanced non-small cell lung cancer in treatment with TKIs and metformin versus TKI alone.

DETAILED DESCRIPTION:
Lung cancer is the first cause of death in men and women, representing 28% and 26% of registered deaths worldwide, respectively. Among patients with this disease, at least 80% has non-small cell lung cancer (NSCLC), and 60% of patients are diagnosed when they already have a locally advanced or metastatic disease. NSCLC therapy regimens depend on the stage of disease and may require surgery, chemotherapy, radiotherapy, or a combination of these. Survival rate at 5 years is low for patients with stage II and III of the disease, with variation from 30% to 5%, this means that an improvement in therapy are required.

Advances in molecular biology of cancer have led to discovering several molecular targets and developing new target therapies. Epidermal growth factor receptor (EGFR) is involved in the development and progression of several types of cancer, including NSCLC. However, despite clinical success with different tyrosine kinase specific domain inhibitors (TKIs), most of the patients respond to these drugs initially, but eventually develop resistance to these drugs after and average period of time of 10 months. Thus, innovative treatment strategies are required urgently to overcome therapeutic resistance to EGFR-TKIs and to improve survival of patients with NSCLC.

Recently, metformin has been associated with reduction in the global risk of incidence and mortality of different types of cancer, due to its anti-tumor properties. In specific types of cancer, retrospective studies have demonstrated a clinical benefit from the use of metformin combined with the treatment of cancer.

Patients with NSCLC with positive EGFR mutations are highly sensible to specific anti-EGFR tyrosine kinase inhibitors, however, most of the patients who initially respond to these target therapies, will present progression of the disease posteriorly during the treatment, this is known as acquired resistance. Acquired resistance to target therapies was first studied in patients with chronic myeloid leukemia with BCR-ABL translocation treated with Imitanib, an inhibitor of aberrant kinase BCR-ABL. Thanks to research, mutations associated with resistance to treatment with TKIs in NSCLC with positive EGFR mutations were discovered. By several studies, additional mutations were found in the kinase domain and in KRAS in those patients with acquired resistance to Gefitinib or Erlotinib. By PCR it was found that 50% of patients with resistance to TKI develop a specific mutation in exon 20 (T790M). However, the mechanism by which the other 50% of patients develop resistance to anti-EGFR TKI is yet unknown. Some studies have found focal amplification of MET proto-oncogen in 22% of the patients with acquired resistance to Gefitinib. The proposed mechanism is that MET amplification promotes resistance by activation of HER3 depending PI3K pathway. Nonetheless, there are few studies with few patients about MET amplification as a resistance mechanism.

On the other hand, there are patients who have this resistance mutation since the first presentation, or de novo. T790M mutation may be present before exposition to TKI and it's generally found with other activating mutations in EGFR (exon 19 deletion and punctual L858R mutation). A response rate of 8% has been reported in those patients treated with gefitinib or erlotinib whose T790M mutation was positive at the time of the diagnosis, with progression-free survival of 2 months and global survival median of 16 months.

Despite the advances in treatment have increased response rate and progression-free survival with anti-EGFR TKI in patients with presence of activating mutations, most of them will develop resistance mutations (T790M) and disease progression. There is no standard treatment in patients who progress from a first generation anti-EGFR TKI, such as erlotinib and gefitinib. Some studies have used afatinib as second line therapy in patients who had progression, finding a benefit in the progression-free survival, disease control rate up until 58% and delay in the development of lung cancer associate symptoms, thus improving quality of life in patients treated with afatinib.

Acquired resistance will develop in a mean time of 9 to 13 months and the 50% to 60% will be secondary to development of T790M resistance mutation.

The molecular mechanisms that generate acquired resistance to anti-EGFR TKI are not completely clear. We know that around 50% of cases are caused by an acquired mutation in the EGFR T790M and a lower percentage by MET oncogene amplification, nevertheless, there are other proposed molecular mechanisms, such as the activation of mesenchymal-epithelial transition. The latter, refers to changes in the phenotype of epithelial cells to cells with mesenchymal cells phenotype, resulting in increase in motility, proliferation and metastasis of tumor cells. It's been proposed that epithelial-mesenchymal (EMT) is associated with sensitivity to chemotherapy and TKI. Finding an effective therapy for patients who develop T790M resistance mutation is required to overcome resistance to first generation anti-EGFR TKI. Afatinib, as a second generation irreversible anti-EGFR TKI, has demonstrated in some studies to have certain effect in patients with resistance, however, the benefit is marginal. Studies have shown that the union of the tyrosine kinase portion of afatinib in patients with resistance mutation, is 100 times less strong that the union in cells with anti-EGFR activating mutations. Pre-clinical studies have demonstrated that inhibition of IL-6 receptor activation and activation of JAK1/STAT3 pathway overcomes resistance and sensitize again those cells with EGFR resistance mutation.

Metformin is a drug that has been used for several years to treat diabetes mellitus and metabolic syndrome, it's generally well tolerated. Several studies since 1910 have suggested that patients with diabetes are at increased risk to develop cancer. The American Diabetes Association and The American Cancer Society have come to a consensus that suggests a clear association for greater risk of cancer incidence in diabetic patients. The tumors that have been studied with more frequency are in: colon, endometrium, rectus and breast. On the other hand, several epidemiologic and cases and control studies have suggested that the use of metformin decreases risk to develop cancer up until 30% with a hazard ratio (HR) of 0.77 (0.64-0.92) and risk of cancer-specific death with a HR of 0.67 (0.53-0.85). Such protective effect has been seen in all kinds of cancer, but has been more studied in breast, gastrointestinal and lung cancer.

The effect of metformin as chemo-prevention is subject to debate, however, there's more information about its use as adjuvant in the treatment of lung cancer, in combination with chemotherapy or target molecular therapy. Pre-clinical studies in mice have demonstrated that use of metformin per os may decrease the necessary dosage of chemotherapy and may prolong tumor remission. Metformin, by inhibiting repairing and anti-apoptosis mechanisms, increases sensitivity to chemotherapy, especially to platinum. Studies that involve metformin, paclitaxel, carboplatin and doxorubicin, have demonstrated to have an effect in tumor regression and prevention of recurrences up until four times the effect of monotherapy in xenograft models in cellular lines of lung and prostate cancer. Retrospective studies have found a benefit in progression-free survival and global survival in diabetic patients with NSCLC, who also are treated with metformin.

T790M mutation and MET amplification are the main resistance mechanisms to anti-EGFR TKI, other mechanisms such as epithelial-mesenchymal transition (EMT) by TGF-β are resistance mechanisms. TGF-β also induces activation of IL-6 and paracrine activation of the receptor (IL-6R) and at the same time the activation of pathway JAK1/STAT3 and cell immortalization. Pre-clinical studies with cellular lines of lung cancer with anti-EGFR acquired-resistance treatment show that metformin prevents transcription of factors that activate epithelial-mesenchymal transition, inhibiting TGF-β, thus, inhibiting IL-6/JAK1/STAT3 pathway, overcoming anti-EGFR TKI resistance in patients with T790M resistance mutation, in vitro and in vivo. A recent study reports that use of metformin in combination with gefitinib may increase efficacy of the latter, showing anti-proliferative and pro-apoptotic effect in cellular lines of NSCLC. Other studies have shown, by Western-blot, a decrease in levels of phosphorylation and activation of growth pathways MAPK, AKT and mTOR with the use of metformin, found in pre-clinical studies. Currently, a phase I/II study is being carried out to determine effective dose, safety and posteriorly the activity of metformin in combination with erlotinib as second line therapy in patients with NSCLC without EGFR mutation.

The main objective of this study is to assess the progression-free survival period in patients with advanced non-small cell lung cancer in treatment with TKIs and metformin versus TKI alone. The secondary objectives are the response rate, global survival, quality of life, safety, as well as determining the alteration of nutrition parameters associated to the combined use of TKIs and metformin.

Besides the secondary objectives, we want to find new candidate markers in the tumor characteristics to predict anti-tumor activity, as well as the search for serum biomarkers; among which we will analyze EGFR mutations (exon 18-21 mutations), IL-6, IGF-1, as well as determination of LKB-1 molecule expression in tumor tissue. We will associate the prognostic and potential role as possible biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC EGFR mutation-positive
* Use of only Metformin as oral hypoglucemic agent
* ECOG-PS 0-2
* Measurable disease
* Life expectancy >12 weeks

Exclusion Criteria:

* Systemic disease
* Patients with TKI treatment longer than 2 months
* History of other neoplasm in the past 5 years
* Breastfeeding women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Start of treatment until 1-year follow-up

SECONDARY OUTCOMES:
Response Rate | 3 month evaluation after start of treatment
  Inflammatory markers (IL-6, IL-12, TNF-alpha)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, MSc, Study Director — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto National de Cancerologia, México, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Data will be uploaded to a repository in an anonimized manner to preserve patient confidentiality.

REFERENCES:
- [Background] Arrieta O, Varela-Santoyo E, Soto-Perez-de-Celis E, Sanchez-Reyes R, De la Torre-Vallejo M, Muniz-Hernandez S, Cardona AF. Metformin use and its effect on survival in diabetic patients with advanced non-small cell lung cancer. BMC Cancer. 2016 Aug 12;16:633. doi: 10.1186/s12885-016-2658-6. PMID 27519177
- [Background] Shigematsu H, Lin L, Takahashi T, Nomura M, Suzuki M, Wistuba II, Fong KM, Lee H, Toyooka S, Shimizu N, Fujisawa T, Feng Z, Roth JA, Herz J, Minna JD, Gazdar AF. Clinical and biological features associated with epidermal growth factor receptor gene mutations in lung cancers. J Natl Cancer Inst. 2005 Mar 2;97(5):339-46. doi: 10.1093/jnci/dji055. PMID 15741570
- [Background] Goodarzi MO, Bryer-Ash M. Metformin revisited: re-evaluation of its properties and role in the pharmacopoeia of modern antidiabetic agents. Diabetes Obes Metab. 2005 Nov;7(6):654-65. doi: 10.1111/j.1463-1326.2004.00448.x. PMID 16219009
- [Background] Shaw RJ, Lamia KA, Vasquez D, Koo SH, Bardeesy N, Depinho RA, Montminy M, Cantley LC. The kinase LKB1 mediates glucose homeostasis in liver and therapeutic effects of metformin. Science. 2005 Dec 9;310(5754):1642-6. doi: 10.1126/science.1120781. Epub 2005 Nov 24. PMID 16308421
- [Background] Morgillo F, Sasso FC, Della Corte CM, Vitagliano D, D'Aiuto E, Troiani T, Martinelli E, De Vita F, Orditura M, De Palma R, Ciardiello F. Synergistic effects of metformin treatment in combination with gefitinib, a selective EGFR tyrosine kinase inhibitor, in LKB1 wild-type NSCLC cell lines. Clin Cancer Res. 2013 Jul 1;19(13):3508-19. doi: 10.1158/1078-0432.CCR-12-2777. Epub 2013 May 21. PMID 23695170
- [Derived] Arrieta O, Barron F, Padilla MS, Aviles-Salas A, Ramirez-Tirado LA, Arguelles Jimenez MJ, Vergara E, Zatarain-Barron ZL, Hernandez-Pedro N, Cardona AF, Cruz-Rico G, Barrios-Bernal P, Yamamoto Ramos M, Rosell R. Effect of Metformin Plus Tyrosine Kinase Inhibitors Compared With Tyrosine Kinase Inhibitors Alone in Patients With Epidermal Growth Factor Receptor-Mutated Lung Adenocarcinoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):e192553. doi: 10.1001/jamaoncol.2019.2553. Epub 2019 Nov 14. PMID 31486833